CLINICAL TRIAL: NCT00405431
Title: Influence of Post-Operative Cyclosporine 0.05% (Restasis) on the Success of Glaucoma Filtering Surgery
Brief Title: Will Restasis Eye Drops Increase Your Chance of Having a Successful Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Marlene Moster, MD, Attending Surgeon, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #03-598
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: glaucoma filtering surgery; restasis; conjunctival inflammation
MeSH Terms: conditions — Glaucoma | interventions — Cyclosporins; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients received restasis eyedrops during 6 month post-operative period
  Interventions: Drug: Restasis
- 2 (Placebo Comparator): Patients receive artificial tears (Endura) during 6 month post-operative period
  Interventions: Drug: Endura (artificial tears)

INTERVENTIONS:
Drug: Restasis — 1 drop in study eye twice a day X 6 months
  Arms: 1
Drug: Endura (artificial tears) — 1 drop in study eye twice a day X 6 months
  Other Names: Endura
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether reducing inflammation of the surface of the eye with topical Restasis after glaucoma surgery will improve surgical outcomes and increase patient comfort.

DETAILED DESCRIPTION:
Continued use of glaucoma drops can alter the outer surface of the eye and result in swelling and irritation, changing the structure of the eye. This structural change has been found to be a significant risk factor for the failure of glaucoma surgery. A comparison of how well patients do after glaucoma surgery depending on whether they use Restasis (the only prescription medication approved by the FDA for treating dry eye) or artificial tears (which can be purchased without a prescription) for 6 months following their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled glaucoma scheduled for filtering surgery

Exclusion Criteria:

* Under 18 years of age
* Unable to understand informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-03; Primary Completion 2005-06 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | 6 months

SECONDARY OUTCOMES:
ocular inflammation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marlene R. Moster, MD, Principal Investigator — Wills Eye Glaucoma Research Center
Locations (1):
- Wills Eye Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
manuscript has been published.

REFERENCES:
- [Result] Fakhraie G, Lopes JF, Spaeth GL, Almodin J, Ichhpujani P, Moster MR. Effects of postoperative cyclosporine ophthalmic emulsion 0.05% (Restasis) following glaucoma surgery. Clin Exp Ophthalmol. 2009 Dec;37(9):842-8. doi: 10.1111/j.1442-9071.2009.02134.x. PMID 20092592